CLINICAL TRIAL: NCT06028048
Title: Protocol of a Randomized Controlled Trial on the Effectiveness and Cost-effectiveness of a Supported Employment Intervention Aimed at Enhancing Work Participation of Unemployed or Work-disabled Cancer Survivors: the PLACES Study
Brief Title: Enhancing Work Participation of Unemployed and Work-Disabled Cancer Survivors
Acronym: PLACES
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Fenna van Ommen, Prof. dr. Angela de Boer, Professor in Chronic Disease and Work Participation at the Faculty of Medicine at Amsterdam UMC., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24535
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Cancer Survivors; Return to Work
Keywords: Cancer survivors; Return to Work; Reintegration; Unemployment
MeSH Terms: interventions — Palliative Care; Employment, Supported

STUDY DESIGN:
Intervention Model Description: A non-blinded RCT will be conducted with a follow-up of 12 months. The study will compare two arms: (1) an intervention group, in which participants will receive the PLACES intervention, and (2) a control group, in which participants will receive CAU. Data on primary (i.e. obtainment of paid employment) and secondary outcomes (e.g. quality of life and self-efficacy regarding RTW) will be gathered at baseline (T0) and after three (T1), six (T2) and twelve months of follow up (T3) using questionnaires .
Who Masked: Outcomes Assessor
Masking Description: The analyses will be performed blinded after one researcher codes the intervention and control group to either 0 or 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLACES intervention (Experimental): Participants in the intervention group will receive the PLACES intervention during 12-months after randomization.
  Interventions: Behavioral: PLACES
- Care as usual (No Intervention): Participants in the control group will receive usual care from the SSA.

INTERVENTIONS:
Behavioral: PLACES — The PLACES intervention is based on eight IPS principles, ensuring competitive employment, client choice, service integration, personalized benefits counseling, rapid job search, systematic development, and individualized support.
  Coaches: Certified IPS coaches receive training from Phrenos IPS knowledge center and Re-turn. Ongoing support includes video lectures, clarifications with researchers, and biannual collective sessions. Coaches, regionally specialized, implement interventions autonomously.
  Intervention Phases:
  1. Intake and Assessment: Participants meet IPS coaches within three days to discuss goals, procedures, and responsibilities, continuing until objectives are met.
  2. Acquisition and Application: Coaches assist job search and placement, aiming for employment within 30 days.
  3. Placement and Support: Coaches offer personalized support, adapting to needs, scheduling meetings based on preferences.
  The intervention ends at 12 months or when goals are achieved.
  Other Names: Individual Placement and Support (IPS); Supported employment
  Arms: PLACES intervention

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of the PLACES intervention on paid employment re-entry in unemployed and work-disabled cancer survivors, compared to CAU.

Secondary Objectives are:

* To evaluate the cost-effectiveness of the PLACES intervention aimed at unemployed or work-disabled cancer survivors.
* To evaluate the effectiveness of the PLACES intervention on time until paid employment, type of employment, change in working hours, quality of life, quality of working life, work ability, and self-efficacy regarding RTW, in unemployed or work-disabled cancer survivors.
* To evaluate the process of conducting the PLACES intervention in terms of recruitment, reach, dose delivered, dose received, fidelity and context.

Participants in the intervention group will receive the PLACES intervention with a maximum duration of 1 year, and participants in the control group will receive CAU.

DETAILED DESCRIPTION:
Participants in the intervention group (n=82) will receive a tailored supported employment intervention, based on the principles of individual placement and support (IPS). This includes support in seeking, returning to and maintaining paid employment. Participants in the control group (n=82) will receive care as usual. All participants will be asked to complete questionnaires, at baseline (T0), and after three (T1), six (T2) and 12 months (T3) follow-up. The primary outcome is obtainment of paid employment. Secondary outcomes are employment status, time until paid employment, change in working hours, importance of work, RTW expectations, work ability, quality of (working) life, and self-efficacy regarding RTW. Process evaluation and cost-effectiveness analysis will be performed.

It is expected that that a significantly higher proportion of participants in the intervention group will obtain paid employment at any point during 12-month follow-up compared to participants in the control group. Additionally, their health, financial situation and quality of life will be improved. If proven effective, the intention is to implement the intervention in usual rehabilitation care.

The study is funded by the Dutch Cancer Society (KWF) and in collaboration with the Netherlands comprehensive cancer organisation (IKNL) and the social security agency (SSA)

ELIGIBILITY:
In order to be eligible for participation, participants must meet all of the following criteria:

1. Of working age (18-65 years);
2. Diagnosed with cancer between 6 months and 10 years ago;
3. Unemployed and either partially or fully work-disabled
4. They have completed their primary treatment (except long-term treatment such as hormone therapy);
5. An approved reintegration trajectory at the SSA;
6. Seeking paid employment and motivated to initiate work promptly.

Cancer survivors who are unable to speak, read or understand the Dutch language and cancer survivors who got diagnosed with basal cell carcinoma will be excluded from participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Paid employment (yes/no) | 12 months
  The primary outcome measure is paid employment (yes/no) at any point during the 1-year-follow-up. Being in paid employment is operationalised as working in a paid job for at least one hour per week as defined by the central statistics office.

SECONDARY OUTCOMES:
Employment status | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  Participants will be ask about their current work situation. A combination of answer options is possible: fulltime, parttime, self-employed, studying, retired, involuntary unemployed, voluntary unemployed, (partially) work-disabled, employed but on sick leave, unemployed and on sick leave, household/caring for others, and 'other'.
Time until paid employment | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  Time until paid employment will be measured as the number of calendar days between randomization and the first day at paid employment. Participants will be asked about the date they started their new job. This can be used to calculate the number of days between randomization and starting in a new job.
Change in working hours | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  For each current work situation (e.g. part-time, voluntary, etc.) participants will be asked about the number of hours per week they work.The answers at different times of follow-up will be used to calculate the change in working hours.
Importance of work | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  Importance of work will be measured by rating the perceived importance of work in one's current situation on a visual analogue scale (VAS) ranging from 1 to 10, with higher scores indicating higher importance of work.
RTW expectations | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  RTW expectation will be measured using a single question asking participants: 'in your estimation, what is the chance you will be at work in 6 months, measured on a 10-point rating scale from 1 (Very little chance) to 5 (very high chance).
Work ability | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  Work ability will be assessed using a single question of the Work Ability Index (WAI), asking participants to estimate their current work ability compared with their lifetime best (0, cannot work at all, to 10, best ever)
Quality of life | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  Quality of life will be assessed with the Short Form-12 (SF-12), which includes the subscales vitality, physical functioning, bodily pain, general health perceptions, physical role functioning. Scores range from 0 to 100, with higher scores indicating higher quality of life.
Quality of working life | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  Quality of working life will be measured with the 23-item cancer-specific quality of working life questionnaire (QWLQ-CS, 23 items). Scores range from 0 to 100 with higher scores indicating a better quality of working life.
Self-efficacy regarding RTW | Baseline (T0), after 3 months (T1), After 6 months (T2) and after 12 months (T3)
  Self-efficacy regarding RTW is measured using the 11-item self-efficacy scale developed by Lagerveld et al. Each item is rated on a 6-point scale and an average score is used to determine the self-efficacy with a higher score (between 1 and 6) indicating better self-efficacy for RTW.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - UWV, Haarlem
  - UWV Zaandam, Zaandam

IPD SHARING:
Plan to Share IPD: Undecided
Questionnaire data will be gathered via Castor EDC (GCP-approved). Amsterdam UMC, location AMC has a processor agreement with Castor EDC: AMC Intranet - Castor EDC. All quantitative data will be stored in Access and SPSS databases. Data will be handled confidentially. Participants' personal data will be pseudonymized by means of codes that do not contain any identifiable information. A participant identification code list will be used to link the data to the participants. The key to the code list will be stored separately from the pseudonymized dataset. The code list will be stored in a locked storage area in the work office and safeguarded by the project leader. Only authorized members of the research team will have access to the key. The pseudonymized dataset will be stored on a secured Amsterdam UMC location AMC server, and safeguarded by authorized members of the research team, for 15 years.

REFERENCES:
- [Derived] van Ommen F, Duijts SFA, Coenen P, Dalton SO, Kliffen A, van Hummel R, de Boer AGEM, Greidanus MA. Protocol of a randomized controlled trial on the effectiveness and cost-effectiveness of the PLACES intervention: a supported employment intervention aimed at enhancing work participation of unemployed and/or work-disabled cancer survivors. Trials. 2024 Sep 9;25(1):603. doi: 10.1186/s13063-024-08441-x. PMID 39252084